CLINICAL TRIAL: NCT05898711
Title: Quality and Safety Outcomes: Prospective Follow Up Registry on FDA Cleared Acellular Fish Skin Grafts in Soft Tissue Reinforcement.
Brief Title: Kerecis Case Registry for SurgiBind : Soft Tissue Reinforcement
Status: Active, not recruiting | Type: Observational
Sponsor: Kerecis Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: KS-0710
Record Dates: First submitted 2023-06-01; First posted 2023-06-12 (Actual); Last update posted 2024-12-31 (Actual); Status verified 2024-10

CONDITIONS: Surgery-Complications

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- All patients: All patients who meet inclusion/exclusion criteria
  Interventions: Device: Fish skin graft

INTERVENTIONS:
Device: Fish skin graft — Kerecis Fish Skin Graft - SurgiBind

SUMMARY:
Registry Objectives The overall objective of the registry is to collect quality and safety data to assess the long-term outcomes of Kerecis Omega3 SurgiBind in surgical procedures to reinforce soft tissue and prevent surgical complications. The ultimate goal of the registry is to enhance the quality of care, patient outcomes and establish a resource to facilitate the use of fish skin in preventing surgical wound dehiscence and surgical site infection.

DETAILED DESCRIPTION:
This Registry is a non-experiment non-interventional case registry to collect quality and safety data on patients that have been treat with the Kerecis product SurgiBind as their regular operative plan from their health care provider.

Primary Objective To collect and quantify patient safety and quality outcomes on a commercially available FDA cleared product Kerecis Omega3 SurgiBind utilized in surgical treatment to reinforce soft tissue and preventing surgical complications (dehiscence and infection).

Secondary Objective To assess the applicable complications post-surgery following the use of fish skin regarding time to heal, time to physical therapy, length of stay, etc.

Registry Procedures Specific Training Prior to patient enrollment, the Sponsor will initiate in person or virtual site visit with participating sites to provide training to the physicians and their staff about the protocol, registry procedures and data entry. The Sponsor will implement a number of strategies to ensure the quality, consistency and interpretability of data recorded. Training, education and ongoing liaison with participating sites will be provided to support high quality data collection.

Recruitment of participants Patients contacting the participating site to schedule the appointment for consultation about their upcoming surgery will be informed about the registry and will be given the option to participate. When the patient comes to the clinic for their visit, information regarding registry participation will be provided by a qualified research staff member. This oral information will be provided while the person is in a private room. Patients can also be recruited through recommendation from their doctors and health care providers.

Data Collection When a subject enrolls in the registry, a unique subject identification number will be assigned. After registry enrollment, data will be collected by the registry physician or trained site personnel either during the routine clinical visit or by telephone contact.

Registry Duration Patients will remain active in the registry for a period of 12 months, no additional information will be collected after that time. Registry enrollment will be for a period of at least 2 years. Registry analysis will be completed in 3 years.

Data Management and Quality Plan Data De-identification Patients enroll in the registry will be assigned a unique subject identification number. This number will consist of ten characters for the registry protocol number, three digits for a site number and four digits for a sequentially assigned subject number (i.e., 0001, 0002, 0003, etc.).

Data Confidentiality, Storage, and Retention All clinicians and related medical staff involved in looking after patients during the study are bound by medical confidentiality and are obliged to comply with data protection follow all Health Information Portability and Accountability Act of 1996 (HIPAA) and Protected Health Information (PHI). Data security is compliance with applicable federal and state laws, rule and regulations, including HIPAA regulation. Research results relating to this study are intended for use in an anonymous form in scientific publications. Personnel who process, generate report or otherwise have contact with PHI must uphold the patient's rights to confidentiality and will be trained in HIPAA privacy and security. If individuals authorized to view records are not bound by medical confidentiality as mentioned above, personal data that come to their attention during checks are confidential under the Data Protection Act.

Data will be collected in a form of case report form (CRF) and entered into secure, web-based portal databases. All users of the databases will need to log in to the databases through a pre-configured username and password controlled by administrator of the system. The databases are housed and managed in an International Organization for Standardization (ISO) 27001 certified environment. Only authorized users and site administrator can see site-wide data. Surgeon Users can only see their procedure. The registry will contain a built-in exporting function to enable data extraction by participating sites to help clinicians review their practice and improve the services. The paper formed CRF will be stored in a locked file cabinet at the participating sites and will be shredded after 7 years post completion of the registry.

Data Quality The registry will implement several strategies to maintain data quality and consistency such as routine cleaning, quality check and periodic feedback. Training, education and ongoing liaison with participating sites will be provided to supporting high quality data collection.

Data Sharing Data can only be shared between participating sites upon request that will be reviewed and approved by the Registry staff. The shared data is only for the purpose of clinical practice improvements, training models and benefiting the patient wellbeing. The registry staff will also provide participating sites with site reports on a regular basis.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion Criteria

  1. Age 18 and older
  2. Undergoing surgical procedure requiring soft tissue reinforcement with Kerecis Omega3 SurgiBind

     For example:
     1. Plastic reconstructive surgery
     2. Orthopedic surgery
     3. Cardiothoracic surgery
     4. Vascular Surgery
     5. General Surgery

     Exclusion Criteria:

  <!-- -->

  1. Participants who request not to be in the registry
  2. Life expectancy of less than 1 year

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients over the age of 18 that are scheduled for surgery and part of their surgical plan is to be treated with Kerecis SurgiBind product for soft tissue reinforcement.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-01-27 (Actual); Primary Completion 2025-06-27 (Estimated); Study Completion 2026-01-27 (Estimated)

PRIMARY OUTCOMES:
Number of surgical complication: dehiscence, infection | 12 months
  quantify the number of patients who experience postoperative wound complications including dehiscence and infection. Patients undergoing surgical procedures and experience wound complications are captured. Wound dehiscence will be categorized as superficial or deep. Infection (if appears) will be identified and recorded. Wounds are considered infected if the wound margins are erythematous and have one or combined of the following: active purulence or necrosis of underlying soft tissues.

SECONDARY OUTCOMES:
Time to healing: | 12 months
  Time to healing: wounds are considered healed when the incision is completely epithelialized with no surrounding erythema
Time to physical therapy initiation | 12 months
  Time it takes for patient to begin physical therapy after the surgical procedure
Duration of physical therapy | 12 months
  How long patient required physical therapy after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Kerecis, Arlington, Virginia, United States